CLINICAL TRIAL: NCT00602329
Title: A Phase II Study Assessing Tumor Blood Flow as Measured by Dynamic Contrast Enhanced MRI in Patients With Metastatic Colorectal Cancer Receiving FOLFOX Alone Versus Patients Randomized to Receive FOLFOX Plus Bevacizumab at 5mg/kg or 10mg/kg.
Brief Title: MRI in Predicting Response in Patients Receiving Combination Chemotherapy and Bevacizumab For Advanced or Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Poor accrual
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000580810; UPCC-09205; GENENTECH-UPCC-09205; UPCC-804021
Record Dates: First submitted 2008-01-19; First posted 2008-01-28 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer; stage III colon cancer; stage III rectal cancer; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (Experimental): Patients receive leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours (FOLFOX) beginning on day 1. Patients also receive bevacizumab at 5 mg/kg IV over 90 minutes on day 1. Treatment repeats every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (Experimental): Patients receive FOLFOX as in arm I and bevacizumab at 10 mg/kg IV over 90 minutes on day 1. Treatment repeats every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin
- FOLFOX alone (control) (Active Comparator): Patients receive FOLFOX as in arm I.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Arms: Arm I; Arm II
Drug: fluorouracil — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving bevacizumab together with combination chemotherapy may kill more tumor cells. Diagnostic procedures, such as MRI, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This randomized phase II trial is studying how well MRI works in predicting response to combination chemotherapy given together with bevacizumab in treating patients with advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the alteration of tumor blood flow using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) in patients with advanced or metastatic colorectal cancer after 2 courses of combination chemotherapy comprising oxaliplatin, fluorouracil, and leucovorin (FOLFOX) and bevacizumab at 5 mg/kg vs 10 mg/kg or FOLFOX alone.

Secondary

* To correlate tumor blood flow, as assessed by DCE-MRI, with time to progression in patients receiving bevacizumab at 5mg/kg vs 10mg/kg.
* To correlate vascular proliferation, as measured by DCE-MRI, with markers of endothelial cell proliferation (i.e., CD31, 34, 105; integrin αvß3; phospho-ERK; Ki67; PCNA; and smooth muscle actin).
* To obtain pilot data on whether assays that measure vascular endothelial cell mitogenic stimulation and mitogenic activity may predict response to therapy, time to progression, and overall survival of patients receiving bevacizumab at 5mg/kg vs 10mg/kg.
* To investigate the association of various markers of apoptosis in tumor cells (e.g., MIF, CREB, or HIF-1-alpha expression/polymorphism and others) and tumor vascularity, as assessed by DCE-MRI.
* To correlate markers of apoptosis in tumor cells with response to therapy, time to progression, and overall survival.
* To determine serum levels of VEGF prior to the initiation of chemotherapy and then prior to courses 2 and 3 of chemotherapy as potential markers of antiangiogenic activity.

OUTLINE: Patients who are eligible to receive bevacizumab are randomized to 1 of 2 treatment arms. Patients who are ineligible to receive bevacizumab receive FOLFOX alone.

* Arm I: Patients receive leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours (FOLFOX) beginning on day 1. Patients also receive bevacizumab at 5 mg/kg IV over 90 minutes on day 1. Treatment repeats every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive FOLFOX as in arm I and bevacizumab at 10 mg/kg IV over 90 minutes on day 1. Treatment repeats every 14 days for 6 months in the absence of disease progression or unacceptable toxicity.
* FOLFOX alone (control): Patients receive FOLFOX as in arm I. All patients undergo dynamic contrast-enhanced MRI at baseline and between courses 2 and 3 (between days 17 and 29) to assess tumor blood flow.

Tumor tissue specimens are obtained from prior colonoscopic biopsy or surgical resection in patients receiving bevacizumab. Tissue specimens are examined by immunohistochemistry to evaluate tumor markers of angiogenesis and apoptosis (e.g., CD31, 34, 105, phospho-ERK, PCNA, Ki67, SMA, and integrin αvß3). Blood specimens are obtained at baseline and prior to courses 2 and 3 (days 15 and 29) to evaluate plasma levels of VEGF.

After completion of study therapy, patients are followed every 2 months for 1 year and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced or metastatic adenocarcinoma of the colon or rectum
* Patients receiving bevacizumab must have tumor tissue available for immunohistochemical analysis

  * Formalin-fixed, paraffin-embedded tissue from previous biopsy or surgical resection is sufficient
* Measurable disease, defined by RECIST as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques (i.e., CT or MRI)

  * CEA elevation alone is insufficient for study entry
* No known brain metastases

PATIENT CHARACTERISTICS:

Criteria for all patients

* ECOG performance status 0-1
* Life expectancy > 3 months
* Granulocytes ≥ 1,500/mL
* Platelet Count ≥ 100,000/mL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST ≤ 5 times ULN
* Urine protein:creatinine ratio ≤ 1.0 at screening
* Patients with other prior malignancies are eligible, provided they have been treated with curative intent and have no evidence of recurrence
* Not pregnant or nursing
* Negative pregnancy test
* No contraindications to MRI, including any of the following:

  * Hypersensitivity to gadolinium
  * Metallic device, including pacemaker, non-MRI compatible aneurysm clip, other non-MRI-compatible mechanical and/or electrical device, or metallic fragments
  * Severe claustrophobia

Additional criteria for patients receiving bevacizumab:

* No significant traumatic injury within the past 28 days
* No serious nonhealing wounds, ulcers, or bone fractures
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No myocardial infarction, unstable angina, or cerebrovascular accident within the past 6 months
* No clinically significant peripheral vascular disease
* No New York Heart Association class II-IV congestive heart failure
* Patients with pre-existing hypertension should be on a stable antihypertensive regimen with blood pressure ≤ 150/100 mm Hg at study entry

PRIOR CONCURRENT THERAPY:

Criteria for all patients

* Prior adjuvant treatment including oxaliplatin allowed
* No prior bevacizumab
* At least 14 days since prior radiotherapy and recovered
* More than 6 months since prior chemotherapy
* No other concurrent investigational agents

Additional criteria for patients receiving bevacizumab:

* At least 28 days since prior major surgical procedure or open biopsy
* At least 7 days since prior minor surgical procedure (e.g., fine-needle aspirations or core biopsies)
* No anticipation of need for a major surgical procedure during study treatment
* Concurrent oral or parenteral anticoagulation therapy allowed provided dose is stable

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-02; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Analysis of tumor blood flow, assessed by DCE-MRI as percentage change in Ktrans, after 2 courses of FOLFOX and bevacizumab or FOLFOX alone compared to baseline value | 2 cycles for all subjects

SECONDARY OUTCOMES:
Analysis of tumor markers of angiogenesis and apoptosis, and the effect of treatment | 2 cycles for all subjects
Correlation of tumor blood flow with time to progression | 2 cycles
Correlation of markers of apoptosis in tumor cells with response to therapy, time to progression, and overall survival | 2 cycles for all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States